## Post Card Consent

Study Title: Invested in Diabetes

Principal Investigator: Bethany Kwan, PhD, MSPH

COMIRB No: 17-2377 Version Date: 3/9/2018

You are being asked to be in this research study because you are a staff member or provider in a practice that is participating in the Invested in Diabetes. Your participation in this portion of the study involves participation in this confidential interview and/or written questionnaire, which should take about up to 60 minutes to complete. There are no costs to you. This research is being paid for by a grant from the Patient Centered Outcomes Research Institute (PCORI).

This study is designed to learn more about different types of shared medical appointments for patients with diabetes. Potential benefits include an improved understanding of how to best help patients with diabetes have as healthy a lifestyle as possible. Practices may learn information they can use to promote more effective implementation of diabetes efforts and improved quality of life for their patients.

The study has minimal risk, limited to the rare but significant risk of loss of confidentiality. Every effort will be made to protect your privacy and confidentiality. Questionnaire and interview data will be completely confidential, and only used by the study team. Data will be reported in aggregate form so that it is not possible to identify you orany individuals. To mitigate potential risks, we will only present results in aggregate at the practice-level, and all data will be stored on a secure research server maintained by the University of Colorado Denver. Data collected will be de-identified as quickly as possible and securely transferred to the University of Colorado. To facilitate the interview today, I would like your permission to record the interview, which will be professionally transcribed. During transcription, all names will be removed and a file number will be placed instead as an identifier.

Your participation in this research is voluntary; you have a choice about being in this study. You do not have to be in this study if you do not want to be. You may choose not to answer certain questions if you are uncomfortable. You may choose to withdraw at any time without penalty. Declining participation will not penalize you in any way from your employment. Your participation or non-participation in this study will not be shared with your employer.

If you have questions, you can call the principal investigator, Dr. Bethany Kwan, at 303-724-5153 or email to <a href="mailto:bethany.kwan@ucdenver.edu">bethany.kwan@ucdenver.edu</a>. If you have questions or concerns about your role and rights as a research participant, would like to obtain information or offer input, or would like to register a complaint about this study, you may contact, anonymously if you wish, the Colorado Multiple Institutional Review Board (COMIRB) at 303-724-1055 or email at COMIRB@ucdenver.edu.

By participating in this interview or the questionnaire, you are agreeing to participate in this research study.